CLINICAL TRIAL: NCT04812158
Title: Effect of Mindfulness Training in Chronic Ankle Instability Among Collegiate Athletes
Brief Title: Video Aided Mindful Deep Breathing for Pain Management
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universiti Tunku Abdul Rahman (Other)
Responsible Party: Principal Investigator, Lee Poh Foong, Assistant professor, Universiti Tunku Abdul Rahman
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Supportive Care
Other Study IDs: VAMDB01; INTI-FHLS-04-01-2016 (Other Grant/Funding Number: INTI INTERNATIONAL UNIVERSITY); EMOTIV, 6251/L29 (Other Grant/Funding Number: University Tunku Abdul Rahman)
Record Dates: First submitted 2021-02-25; First posted 2021-03-23 (Actual); Last update posted 2021-03-23 (Actual); Status verified 2021-03

CONDITIONS: Musculoskeletal Pain; Ankle Injuries; Joint Instability
Keywords: Mindfulness; Breathing; Rehabilitation; Athletes; Physiotherapy; Electroencephalography
MeSH Terms: conditions — Musculoskeletal Pain; Ankle Injuries; Joint Instability; Respiratory Aspiration | interventions — Rehabilitation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control group (Active Comparator): participants in the control group receive gold standard physiotherapy intervention 5 times a week for 6 weeks
  Interventions: Other: standard ankle physiotherapy or rehabilitation for chronic ankle instability
- Experimental group (Experimental): 3 min video-aided mindful deep breathing (VAMDB) or visual guiding on deep breathing with 6 deep breath per minute along with standard physiotherapy (SP) protocol and the control group was given standard physiotherapy (SP) protocol 5 times a week for 6 weeks
  Interventions: Other: standard ankle physiotherapy or rehabilitation for chronic ankle instability
- Healthy control (No Intervention): Active healthy participants who engaged in regular collegial sports

INTERVENTIONS:
Other: standard ankle physiotherapy or rehabilitation for chronic ankle instability — 6 weeks of combined interventions of video aided mindful deep breathing and standard ankle physiotherapy in rehabilitating the chronic ankle instability for participants with chronic ankle instability
  Other Names: Video aided mindful deep breathing with standard ankle physiotherapy or rehabilitation for chronic ankle instability
  Arms: Control group; Experimental group

SUMMARY:
Chronic ankle instability (CAI) is the most common musculoskeletal injury in sports and the rate of CAI accounts for 85% of ankle injuries. It has been estimated that 23,000 ankle sprains occur each day in the United States, representing approximately 1 sprain per 10,000 people per day and nearly one in five ankle injuries result in chronic symptoms. Numerous researchers applied mindfulness for improving the performance of various sports such as table tennis, shooting, cricket, archery, golf, swimming, and cycling. Since many of the players do not possess effective pain coping skills, they are at risk for lifelong impairment of their emotional, social, and physical functioning. Mindfulness-centered interventions may well serve to mitigate pain-related disability. Training in mindfulness meditation improves anxiety, depression, stress, and cognition. Mindfulness-related health benefits are associated with enhancements in cognitive control, emotion regulation, positive mood, and acceptance, each of which have been associated with pain modulation. Since mindfulness has been proven effective in managing various health disorders and in enhancing sports performance, our study aims to apply the mindfulness approach in rehabilitating the most common sports injury, CAI. The improvement in CAI due to the mindfulness approach will be assessed by the improvement in pain response through the Cumberland ankle instability tool, Functional ankle disability index (FADI), Visual analog scale (VAS), Brief Pain Inventory (BPI), Y-balance test, Mindfulness attention awareness score (MAAS), Oxford Happiness Questionnaire (OHQ) quantitative electroencephalography (Q-EEG). This study finding will be useful in assessing the effectiveness of mindfulness in rehabilitating CAI and identify the correlation of CAI pain response with VAS & BPI, quantitative electroencephalography - Q-EEG. In this clinical trial, the investigators wish to use noninvasive methods such as quantitative EEG (electroencephalogram) to find the brainwave patterns during the different stages of mindfulness intervention (pre and post). The outcome of this study will eventually lead to the identification of a better assessment method to indicate the pain response for the appropriate physiotherapy management. The application of mindfulness technique in CAI management and the usage of Q- EEG to assess the pain response in chronic ankle injury athletes are the novel approaches of this research study.

DETAILED DESCRIPTION:
Background:

Inversion Ankle injuries (IAS) are among the most common musculoskeletal injuries in sports and the rate of IAS accounts for 85% of ankle injuries. The hallmarks of chronic ankle instability (CAI) include repeated ankle sprains that have led to an altered patient activity level. Important factors include injuries sustained, frequency of events, localization of pain, and prior treatment modalities. The degree of disability appreciated by the patient is one of the most important factors and can be significant in both high- and low-demand individuals. The most commonly cited characteristics of CAI include giving way to the ankle, mechanical instability, pain and swelling, loss of strength, recurrent sprain, and functional instability. Residual problems can persist for decades, with up to 72% of people unable to return to their previous level of activity, such as fear of the ankle giving way. Functional ankle instability includes a perceived or actual giving way of the ankle (or both) and other characteristics previously associated with CAI in general: pain, swelling, and recurrent sprain. Functional insufficiencies among individuals with either CAI have been demonstrated by quantifying deficits in ankle neuromuscular response times, postural control, and strength.

Researchers have found that injured athletes experience clinically significant depression 6 times as often as non-injured athletes. Injured athletes also exhibit significantly greater anxiety and lower self-esteem than non-injured. Athletes with more severe injuries are more likely to become depressed than the non-injured. Since many of the players do not possess effective pain coping skills, they are at risk for lifelong impairment of their emotional, social, and physical functioning. Mindfulness-centered interventions may well serve to mitigate a pain-related disability. Training in mindfulness meditation improves anxiety, depression, stress, and cognition. Mindfulness-related health benefits are associated with enhancements in cognitive control, emotion regulation, positive mood, and acceptance, happiness each of which have been associated with pain modulation. Successively mindfulness has been proven effective in managing various health disorders and in enhancing sports performance. This study aims to apply the video-assisted mindfulness deep breathing training (VAMDBT) approach in rehabilitating CAI, the most common sports injury. In addition, applies Quantitative Electroencephalogram (QEEG) as one of the parameters to measure the pain response of collegiate athletes.

Literature Chronic ankle pain can affect all age groups, ranging from young athletes to elderly patients with degenerative joint and soft-tissue disorders. Although physical activity brings a range of lifelong health benefits, it may also lead to injuries that pose a significant threat to health. Among 90 Plus League volleyball players age 18-37, over 87% of the respondents suffered from at least one sport-related injury. In total, 362 injuries occurred, on average 4.02 injuries per one volleyball player. The most commonly involved sports injuries were ankle sprains (46 injuries), knee and lower leg muscles (30), interphalangeal articulations of fingers (30) as well as the shoulder joint. More than half of the injuries (57%) occurred twice or three times.

The pattern of musculoskeletal injuries sustained by Malaysian badminton players who attended the National Sports Institute (NSI) Clinic, Kuala Lumpur, Malaysia. The mean age of the players who attended the clinic was 19.2 (range 13-52) years. Approximately 60 percent of the injuries occurred in players younger than 20 years of age. The majority of injuries (91.5 percent) were categorized as mild overuse injuries and mostly involved the knee and ankle. The prevalence of sports injuries among 475 male professional athletes participating in ball sports who are aged 15 years and older, from 5 sports clubs in Kuwait. About 452 athletes from four ball games (football (soccer), basketball, handball, and volleyball) were included in this study. The study found that the overall 12-month and lifetime prevalence of sports injuries were 73.8 and 89.8%, respectively. Lower limbs (73.1%) were the most common site of injuries and joint injuries (43.6%) were the most common type of injury reported. The study analyzed the characteristics of injuries and associated personal and training characteristics in young basketball players of both sexes. A conducted one-year retrospective cross-sectional survey with 581 basketball players (350 males and 231 females) participated in the school games and high school Olympics in the state of São Paulo, Brazil. The study used a questionnaire that contained items addressing anthropometric data and characteristics of injuries that have occurred in the previous 12 months. Results showed a total of 167 of the athletes reported injuries and the male gender exhibited a greater risk of injury than the female gender. The most affected anatomic sites were the ankle/foot and knee. A study that investigates the pattern of muscle injuries and the factors that predict the return-to-play duration among Malaysian athletes who attended the National Sports Institute Clinic. About 397 muscle injuries were diagnosed among 360 athletes from the period June 2006 to December 2009. The median age of the athletes with muscle injuries was 20.0 years. Muscle injuries were mostly diagnosed among national-level athletes and frequently involved the lower limb. There is a twofold increased risk for ankle injury recurrence for at least one-year post-injury. In up to 50% of all cases, recurrences result in disability and lead to chronic pain or instability, requiring prolonged medical care. Therefore, ankle sprain recurrence prevention in athletes is essential. A study that measured preseason anxiety and depression reported a total of 597 injuries with 40.6% preseason injuries, 28.8%, and 21.7% of athletes suffered from anxiety and depressive symptoms. Another study stated depression and anxiety disorders have a negative effect on subjective well-being. The Oxford Happiness Scale, Life Satisfaction Scale response among 284 patients shows that participants were found to be moderately happy and satisfied.

Chronic Ankle Injury Rehabilitation Ankle sprains are a common problem seen by primary care physicians, especially among teenagers and young adults. Early mobilization speeds healing and reduce pain more effectively than prolonged rest. A previous ankle sprain is the greatest risk factor for an acute ankle sprain, it is important to counsel the recovering patients on prevention strategies. Ankle braces and supports, ankle taping, a focused neuromuscular training program, and regular sport-specific warm-up exercises have proven to protect against ankle injuries, and have to be considered for patients returning to sports or other high-risk activities.

Mindfulness Recent attention in healthcare research has been paid to the concept of mindfulness and its contributions to clinical practice. Mindfulness refers to the way individuals pay attention to their experiences from moment to moment with non-judgmental attitudes. The cultivation of mindfulness requires regular practice of mindful breathing and different types of meditation. Mindfulness meditation has been found to improve a wide spectrum of cognitive and health outcomes. Training in mindfulness meditation improves anxiety, depression, stress, and cognition. Mindfulness-related health benefits are associated with enhancements in cognitive control, emotion regulation, positive mood, and acceptance, each of which has been associated with pain modulation. Thus, it seems reasonable to hypothesize that mindfulness meditation itself would attenuate pain through some of these mechanisms. A mindfulness training for eight weeks duration was shown to improve pain acceptance in lower back pain patients. Neurophysiological changes are consistent with a bio-psycho-social formulation reflecting the underlying mechanisms associated with sensory and motor findings, psychological traits, and perceptual changes associated with chronic musculoskeletal conditions. These changes, therefore, have important implications in the clinical manifestation, pathophysiology, and rehabilitative treatment of chronic musculoskeletal disorders. Musculoskeletal rehabilitation professionals have at their disposal tools to address these neuroplastic changes including top-down cognitive-based interventions (such as education, cognitive behavioral therapy, mindfulness meditation, and motor imagery), and bottom-up physical interventions (such as motor learning, peripheral sensory stimulation, and manual therapy) that induce neuroplastic changes across distributed areas of the nervous system and impact outcomes in patients with chronic musculoskeletal disorders. Mindful exercise executed with profound and nonjudgmental attention to breathing and proprioceptive awareness of muscles and movements.

Assessment of Mindfulness Approach:

A pilot study using an 8-week mindfulness-based stress reduction (MBSR) program on a sample of low back pain patients was conducted in order to assess the feasibility and effectiveness of the intervention as well as changes in an EEG pattern called thalamocortical dysrhythmia which is associated with chronic pain. The study involved 22 patients with chronic low back pain who participated in an MBSR program. The result showed a medium-sized effect for psychological functioning, pain severity, and quality of life. However, EEG analyses revealed no differences between the pre-and post-intervention. The major concerns from the previous mindfulness studies about the participant's compliance reported were time constraints and personal commitments. The high demand in time and the need for guidance from a coach can discourage the community from taking up these practices as well. For a full MBSR course, it can take up to eight weeks, with weekly meetings that last for about three hours and the daily practice of about an hour. This can be difficult to adhere to especially in the current fast-paced lifestyle of young people. With due consideration of participants' compliance, the mindfulness intervention practice of the present study has been modified to 5- min video-assisted mindfulness deep breathing. Furthermore, the follow-up of participants' home practices will be monitored with the use of a smartphone app that has the facility to send reminders as text messages to fill in the practice diaries or online portals to record the frequency of home practice of our intervention. A recent study on short-duration, video-assisted deep breathing among healthy young adults showed that the participants engaged for 5 min deep breathing revealed profound NoGo N2 amplitude increment as compared to the control group in the follow-up session. Results indicated the possibility of performing short-duration deep breathing guided by video-assisted deep breathing to achieve an enhanced conflict monitoring as an alternative to other mindfulness practices. Therefore the objective of this study is to find the effectiveness of VAMDBT in the recovery of chronic ankle instability among collegiate athletes.

ELIGIBILITY:
Inclusion Criteria:

* CAIT scores ≤27
* age ranging from 18 to 25
* male participants
* previous history of ankle sprains
* referred chronic ankle instability for physiotherapy

Exclusion Criteria:

* history of previous surgery
* under pain-relieving medicine
* under deep breathing or meditation
* bilateral ankle sprains
* acute musculoskeletal injuries of lower limb

Ages: 18 Years to 25 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — The brain signals response differs between the genders and the relative power of beta and theta waves found to be dominant in males
Enrollment: 45 (Actual)
Dates: Start 2018-01-15 (Actual); Primary Completion 2019-02-19 (Actual); Study Completion 2019-02-19 (Actual)

PRIMARY OUTCOMES:
Change from baseline ankle stability by Cumberland Ankle Instability Tool (CAIT), 9-item scores at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  Cumberland Ankle Instability Tool (CAIT), is a reliable and valid tool to assess the balance of participants with ≤27 in the CAIT tool over 30, where lower scores represent "poor" ankle stability and higher scores represent "better" ankle stability. Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline dynamic ankle stability by Y-balance test (YBT) scores at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  Y balance test (YBT) is a valid and reliable tool to measure participants' dynamic balance of affected ankle distance in anterior, posterolateral, and posteromedial directions, where lower scores represent "poor" ankle stability and higher scores represent "better" ankle stability. Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline in pain by visual analog scale (VAS) at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  A visual analog scale (VAS) is a valid and reliable self-reported tool to record participants' pain intensity on a 10 cm line to point out the pain level. The point at 0 cm represents "no pain" and 10 cm represents "worst pain", where higher scores represent better ankle stability. Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline in pain by Brief Pain Inventory (BPI) at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  Brief Pain Inventory (BPI) is a valid and reliable tool to record participants pain intensity and interference with the 4- items (worst pain, least pain, average pain, and pain right now) to measure the pain intensity, and 7 -items (general activity, mood, walking, normal work, relations, sleep, enjoyment of life) to assess the pain interference. The participants are instructed to report the pain intensity from 0 (no pain) to 10 (as pain bad as the participants can imagine). Similarly, the pain interference is recorded from 0 (does not interfere) to 10 (completely interferes). Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline ankle stability by Functional ankle disability index (FADI ), 34-item scores at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  Functional ankle disability index (FADI) is a validated tool to assess participant's balance during general daily activity and sports-specific functions, where lower scores represent "poor" ankle stability and higher scores represent "better" ankle stability. Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline attention by Mindful Attention Awareness Scale (MAAS), 15-item scores at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The changes in the mind adaptation of participants are obtained from the Likert scale rating from 1(almost always) to 6 (almost never), MAAS is a reliable tool. Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline attention by Oxford Happiness Questionnaire (OHQ), 29-item scores at week 3, week 6 and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The participants' happiness level is assessed using the reliable tool Oxford Happiness Questionnaire (OHQ), which consists of a 29-item questionnaire. The OHQ score will be recorded on 6 points Likert scale from 1 (strongly disagree) to 6 (strongly agree).
  Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)

SECONDARY OUTCOMES:
Change from baseline Alpha waves by Non-invasive wireless electroencephalogram (EEG) at week 3, week 6, and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The 14- channel electrodes were placed at a sampling rate of 128 Hz, in compliance with the International 10-20 System nomenclature. The increase or decrease in alpha wave EEG recordings of the participants are recorded in eyes closed and eyes open for 2mins.
  Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline Beta waves by Non-invasive wireless electroencephalogram (EEG) at week 3, week 6, and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The 14- channel electrodes were placed at a sampling rate of 128 Hz, in compliance with the International 10-20 System nomenclature. The increase or decrease in beta wave EEG recordings of the participants are recorded in eyes closed and eyes open for 2mins.
  Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline Theta waves by Non-invasive wireless electroencephalogram (EEG) at week 3, week 6, and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The 14- channel electrodes were placed at a sampling rate of 128 Hz, in compliance with the International 10-20 System nomenclature. The increase or decrease in theta wave EEG recordings of the participants are recorded in eyes closed and eyes open for 2mins.
  Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline delta waves by Non-invasive wireless electroencephalogram (EEG) at week 3, week 6, and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The 14- channel electrodes were placed at a sampling rate of 128 Hz, in compliance with the International 10-20 System nomenclature. The increase or decrease in delta wave EEG recordings of the participants are recorded in eyes closed and eyes open for 2mins.
  Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)
Change from baseline gamma waves by Non-invasive wireless electroencephalogram (EEG) at week 3, week 6, and week 12 | Baseline, 3 Weeks,6 Weeks, 12 Weeks
  The 14- channel electrodes were placed at a sampling rate of 128 Hz, in compliance with the International 10-20 System nomenclature. The increase or decrease in gamma wave EEG recordings of the participants are recorded in eyes closed and eyes open for 2mins.
  Change =(Week 3 score - Baseline, Week 6 score - Baseline, Week 12 score - Baseline)

CONTACTS AND LOCATIONS:
Locations (1):
- INTI physiotherapy centre, Nilai, Seremban, Negeri Sembilan, Malaysia

IPD SHARING:
Plan to Share IPD: No
Based on informed consent participants data not shared

REFERENCES:
- [Derived] Ramalingam V, Cheong SK, Lee PF. Effect of six-week short-duration deep breathing on young adults with chronic ankle instability-a pilot randomized control trial. BMC Sports Sci Med Rehabil. 2023 Nov 15;15(1):155. doi: 10.1186/s13102-023-00758-5. PMID 37968738

DOCUMENTS (1):
  • Study Protocol (2018-01-15): https://cdn.clinicaltrials.gov/large-docs/58/NCT04812158/Prot_000.pdf